CLINICAL TRIAL: NCT04322812
Title: Evaluation of the Effects of Photobiomodulation Therapy (PBMT) Combined With Static Magnetic Field (sMF) on Temporary Pain Relief in Fibromyalgia Patients: a Randomized Placebo-controlled Trial
Brief Title: Effects of Photobiomodulation Therapy Combined With Static Magnetic Field in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Multi Radiance Medical (Industry)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2.732.062
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Fibromyalgia
Keywords: Photobiomodulation Therapy; Low-level Laser Therapy; Fibromyalgia; Pain intensity
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A researcher will program the device (placebo or PMBT) and will be instructed not to inform the patients or other researchers as to the type of treatment (PMBT or placebo). Therefore, the researcher responsible for the treatment, the investigator and the outcome assessor will be blinded to the type of treatment being administered to the patients. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (placebo or PBMT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active PBMT (Active Comparator): Active PBMT applied three times a week (interval of 48 hours approximately), for three consecutive weeks, totalling nine treatment sessions.
  Interventions: Device: Active PBMT
- Placebo PBMT (Placebo Comparator): Placebo PBMT applied three times a week (interval of 48 hours approximately), for three consecutive weeks, totalling nine treatment sessions.
  Interventions: Device: Placebo PBMT

INTERVENTIONS:
Device: Active PBMT — The Active PBMT will be applied using MR5™ ACTIV PRO LaserShower Laser Therapy System, manufactured by Multi Radiance Medical (Solon, OH, USA) will be used. The ACTIV PRO emits 30mW of 905nm, 300mW of 850nm, 200mW of 660nm and 0mW of 455nm light via an electric diode energy source. PBMT will be applied using the direct contact method with light pressure on the skin. The PBMT application time will be 120 seconds per region and the total time will vary according to the number of regions to be treated. Only the painful regions on that day will be treated (according widespread pain index [WPI] ), which can comprise a minimum of 3 and a maximum of 18 regions in total. The dose used for applications during the treatment will be 60 Joules (J) per region. The total dose might vary between patients and each session.
  Arms: Active PBMT
Device: Placebo PBMT — The placebo PBMT will be applied using MR5™ ACTIV PRO LaserShower Laser Therapy System, manufactured by Multi Radiance Medical (Solon, OH, USA). The ACTIV PRO emits 905nm, and 850nm via an electric diode energy source with outputs to 0%. The 660nm light via an electric diode energy source with outputs to >1% to appear like the active comparator. PBMT will be applied using the direct contact method with light pressure on the skin. The placebo PBMT application time will be 115 seconds per region and the total time will vary according to the number of regions to be treated. Only the painful regions on that day will be treated (according WPI), which can comprise a minimum of 3 and a maximum of 18 regions in total. The dose used for applications during the treatment will be 0 Joules (J) per region. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (active or placebo).
  Arms: Placebo PBMT

SUMMARY:
Fibromyalgia (FM) syndrome is defined by the American College of Rheumatology (ACR), as a chronic widespread pain and tenderness in at least eleven of eighteen specific tender points. Despite the increased understanding about FM, there is currently no cure for this syndrome and the treatment aims to provide symptomatic relief and improvement of physical capacities to perform daily tasks and quality of life. Evidence has suggest that photobiomodulation therapy (PBMT) can be used as monotherapy or as a supplementary treatment to other therapeutic procedures in patients with FM. However, the lack of consensus regarding therapeutic protocols hinders multicenter comparisons of the many clinical trials published. Further studies are needed to establish ideal parameters of PBMT to be used as a therapeutic tool in the management of fibromyalgia. Therefore, the aim of this project is to investigate the effectiveness of PBMT combined with static magnetic fields (sMF) in pain relief in patients with fibromyalgia.

DETAILED DESCRIPTION:
To achieve the proposed objectives it will be performed a randomized, triple-blind, placebo-controlled trial, with voluntary patients with fibromyalgia. Ninety patients will be randomly allocated to two treatment groups: 1. Active PBMT (MR5™ ACTIV PRO LaserShower) or Placebo PBMT (MR5™ ACTIV PRO LaserShower). The patients will be treated by a blinded therapist.

The patients randomly allocated to the different groups will be subjected to treatment 3 times a week, total of 9 sessions (with approximately 48 hours between each session), a total of 3 weeks of treatment.

The clinical outcomes will be obtained at the stabilization phase, baseline, end of treatment and 30 days after the conclusion of treatment.

The data will be collected by a blinded assessor.

Statistical analyzis:

* The primary statistical method to analyze the primary endpoint will be Fisher's Exact Test to compare the proportion of success between the test (Active PBMT) and the control procedure (Placebo PBMT) groups, considering that randomization has been diligently conducted and important covariates between the two groups are well balanced. Statistical significance is set at p < 0.05.
* Unpaired T test will be applied to analyze pain intensity through EVA. Mean and individual subject changes in VAS ratings across and between all study evaluation time-points, within and between procedure groups considering that randomization has been diligently conducted and important covariates between the two groups are well balanced. Statistical significance is set at p<0.05.
* For patient satisfaction, measured through a Likert Scale, the data will be reduced to the nominal level by combining all agree and disagree responses into two categories of "accept" and "reject". Differences in satisfaction with Study Outcome Ratings between procedure groups at both evaluated time-points, and any change between. The chi-square, will be used after this transformation. Statistical significance is set at p<0.05.

The investigators will analyze: degree of pain rating (tender point count), pain intensity, patient satisfaction and adverse events

ELIGIBILITY:
Inclusion Criteria:

* being female;
* age between 30 and 55 years;
* have an ovulatory cycle;
* height between 1.50m and 1.80m, body mass between 50 and 80 kg and BMI in the range of > or = to 18.5 kg/ m2;
* present a diagnosis of fibromyalgia and meet the current criteria of the American College of Rheumatology;
* had symptoms of fibromyalgia greater than 3 months;
* Widespread Pain Index (WPI) score > or = to 9, Visual Analogue Scale score > or = to 50 Fibromyalgia Impact Questionnaire score > or = to 50
* is not pregnant;
* not having diabetes mellitus and uncontrolled blood pressure;
* not having psychiatric illness or having malignant tumors;
* did not present dengue, Zika or Chikungunya in the last year;
* not to be hypersensitive to light;
* cognitive level enough to understand the procedures and follow the guidelines;
* consent to participate in the study and sign the consent form.

Exclusion Criteria:

* arthritis, chronic fatigue syndrome, lupus, auto-immune diseases;
* cognitive changes;
* people who perform some exercise;
* having a pacemaker;
* people under the age of 30 and more than 55 years;
* injuries in the last 6 months;
* not attend for more than two consecutive sessions;
* at any time and for any reason expressing an intention to leave the study.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Degree of pain rating - change of TCP (tender point count) | 3 weeks (end of treatment) and 4 weeks after the conclusion of the treatment.
  Reduction of the tender point count (TCP) where they have experienced pain as reported on Fibromyalgia Impact Questionnaire (FIQ).

SECONDARY OUTCOMES:
Pain intensity - VAS | 3 weeks (end of treatment) and 4 weeks after the conclusion of the treatment.
  Pain intensity will be measured by 0-100 standardized Visual Analog Scale (VAS).
Patient satisfaction - Likert Scale | 3 weeks (end of treatment) and 4 weeks after the conclusion of the treatment.
  Patient satisfaction will be measured by 1-item Likert Scale. The scale uses the following responses: very satisfied = 4; somewhat satisfied = 3; not very satisfied = 2; not at all satisfied =1. Highest scores indicates better satisfaction.
Adverse events | 3 weeks (end of treatment) and 4 weeks after the conclusion of the treatment.
  Adverse events will be measured by report.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Cesar Pinto Leal Junior, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Laboratory of Phototherapy and Innovative Technologies in Health, São Paulo, Brazil